CLINICAL TRIAL: NCT05267054
Title: A Phase 1b/2 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of Ociperlimab (BGB-A1217) in Combination With Tislelizumab (BGB-A317) or Rituximab in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: Treatment of Relapsed or Refractory Diffuse Large B Cell Lymphoma With Ociperlimab (BGB-A1217) in Combination With Tislelizumab (BGB-A317) or Rituximab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdvanTIG-101; CTR20220360 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-02-10; First posted 2022-03-04 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma; Refractory Diffuse Large B-cell Lymphoma
Keywords: Lymphoma; Tumor; Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Neoplasms | interventions — tislelizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ociperlimab + Tislelizumab (Experimental): Participants received ociperlimab 900 mg and tislelizumab 200 mg every three weeks (Q3W) by intravenous injection (IV) until confirmed progressive disease, death, withdrawal of consent, loss of follow-up, or the end of study.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab
- Ociperlimab + Rituximab (Experimental): Participants received ociperlimab 900 mg and rituximab 375 mg/m² Q3W by intravenous injection until confirmed progressive disease, death, withdrawal of consent, loss of follow-up, or the end of study.
  Interventions: Drug: Ociperlimab; Drug: Rituximab

INTERVENTIONS:
Drug: Ociperlimab — administered intravenously
  Other Names: BGB-A1217
Drug: Tislelizumab — Administered intravenously once every 3 weeks
  Other Names: BGB-A317; Tevimbra
  Arms: Ociperlimab + Tislelizumab
Drug: Rituximab — Administered intravenously once every 3 weeks
  Arms: Ociperlimab + Rituximab

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of ociperlimab (BGB-A1217) in combination with tislelizumab (BGB-A317) or rituximab in participants with relapsed or refractory (R/R) diffuse large B cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed DLBCL NOS (Not Otherwise Specified), Epstein-Barr virus (EBV) + DLBCL NOS, or high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (double/triple-hit lymphoma [DHL/THL]), based on the World Health Organization (WHO) 2016 classification of tumors of hematopoietic and lymphoid tissue

   1. Cohort 1: participants must have positive tumor programmed cell death ligand-1 (PD-L1) immunohistochemistry (IHC) testing results as determined by local pathologist
   2. Cohort 2: Participants must have negative tumor PD-L1 IHC results as determined by a local pathologist in the dose confirmation stage. The dose expansion stage can enroll participants regardless of PD-L1 expression.
2. Previously received ≥ 1 line of adequate systemic anti DLBCL therapy, defined as an anti CD20 antibody based chemoimmunotherapy for ≥ 2 consecutive cycles, unless participants had PD before Cycle 2.
3. Relapsed or refractory disease before study entry, defined as either:

   1. Recurrent disease after having achieved disease remission (complete response or partial response) during or at the completion of the latest treatment regimen.
   2. Stable disease or progressive disease (PD) at the completion of the latest treatment regimen.
4. Ineligible for high dose therapy/hematopoietic stem cell transplantation
5. Measurable disease as assessed by computed tomography (CT) or magnetic resonance imaging (MRI) and defined as at least 1 lymph node > 1.5 cm in the longest diameter and/or at least 1 extranodal lesion > 1.0 cm in the longest diameter, and measurable lesion (s) in 2 perpendicular diameters

Exclusion Criteria:

1. Current or history of central nervous system lymphoma
2. Histologically transformed lymphoma
3. Receipt of the following treatment:

   1. Systemic chemotherapy, targeted small molecule therapy or radiation therapy within 4 weeks (or 5 half lives, whichever is shorter) before first dose of study drug
   2. Recent treatment with another monoclonal antibody within 4 weeks before first dose of study drug
   3. Investigational treatment within 4 weeks (or 5 half lives, whichever is shorter) before first dose of study drug
   4. Treatment with autologous stem cell transplantation within 6 months before first dose of study drug
   5. Treatment with allogeneic hematopoietic stem cell transplantation or organ transplantation
   6. Treatment with anti-programmed cell death protein-1 (PD-1), anti PD-L1, anti PD-L2, anti T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif (ITIM) domain (TIGIT), anti CTLA4 or other antibody or drug specifically targeting T cell costimulation or checkpoint pathways.
4. Active autoimmune diseases or history of autoimmune diseases that may relapse, with the following exceptions:

   1. Controlled Type 1 diabetes
   2. Hypothyroidism (provided that it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, or alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began in April 2022 and completed in August 2024. Fifty-three participants were enrolled in this study, and all received treatment.
Groups:
- Ociperlimab + Rituximab: Participants received ociperlimab 900 mg and rituximab 375 mg/m^2 Q3W by intravenous injection until confirmed progressive disease, death, withdrawal of consent, loss of follow-up, or the end of study.
Period: Overall Study
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Started | 24 | 29
Completed | 0 | 0
Not Completed | 24 | 29
Not completed — Death | 13 | 14
Not completed — Study Ended by Sponsor | 9 | 13
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Median (Full Range); unit: Years] — Baseline is defined as last non-missing value collected before the first dose of study drug.
  Years | 64.0 [40 to 79] | 66.0 [21 to 80] | 65.0 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 10 | 16 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 24 | 29 | 53
Region of Enrollment [Number; unit: participants]
  China | 24 | 29 | 53
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Scale is used to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature
  2. = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours
  4. = Completely disabled, confined to bed or chair
  5. = Dead
  Participants
    Grade 0 | 8 | 8 | 16
    Grade 1 | 16 | 21 | 37
    Grade 2 | 0 | 0 | 0
Weight [Median (Full Range); unit: kg] | 59.00 [45.5 to 102.0] | 63.80 [45.0 to 90.0] | 62.00 [45.0 to 102.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug(s), whether considered related to study drug(s) or not.
  An SAE is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the investigator based on medical judgement (eg, may jeopardize the patient or may require medical/surgical intervention to prevent one of the outcomes listed above).
Time Frame: From first dose of study drug up to 30 days after last dose, maximum time on treatment was 98 weeks.
Population: The Safety Analysis Set is defined as all participants who received any dose of any study drug(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 24 | 29
Participants
  Treatment Emergent Adverse Events | 24 | 28
  Serious Adverse Events | 9 | 8

2. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Ociperlimab When Administered in Combination With Tislelizumab or Rituximab
Description: The highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 33.3%
Time Frame: 21 days
Population: Safety analysis set
Measure: Number; unit: mg Q3W
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 24 | 29
mg Q3W | 900 | 900

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best overall response of partial response (PR) or complete response (CR) based on the Lugano classification as assessed by the investigator. Response was evaluated using computed tomography (CT) and metabolic imaging (fluorodeoxyglucose-positron emission tomography (FDGPET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  PR is partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
Time Frame: From first dose of study drug to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy Analysis Set is defined as all the participants who received any dose of any study drug(s), had evaluable disease at baseline, and had at least one evaluable post-baseline tumor assessment unless clinical progression or death occurred prior to first tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 23 | 27
percentage of participants | 17.4 [5.0 to 38.8] | 18.5 [6.3 to 38.1]

4. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants who achieved a complete response per the Lugano Classification (2014) as assessed by the investigator.
Time Frame: From first dose of study drug to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 23 | 27
percentage of participants | 13.0 [2.8 to 33.6] | 7.4 [0.9 to 24.3]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date that response criteria were first met to the date that progressive disease is objectively documented per Lugano Classification (2014), as assessed by the investigator, or death, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: Up to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy analysis set; participants with a best overall response of CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 4 | 5
Months | 13.34 [6.2 to 18.7] | 7.82 [0.0 to 8.5]

6. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from study treatment start to date of the earliest qualifying response (partial response or better) per Lugano Classification (2014) as assessed by the investigator
Time Frame: From first dose of study drug to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy analysis set; participants with a best overall response of CR or PR.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 4 | 5
months | 2.09 [2.07 to 2.17] | 2.04 [1.97 to 2.40]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose until first documentation of progression per Lugano Classification (2014), as assessed by the investigator, or death, whichever comes first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From first dose of study drug to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 23 | 27
Months | 1.2 [0.9 to 1.9] | 1.8 [0.9 to 2.2]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first study drug administration to the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From first dose of study drug to the data cutoff date of 30 August 2024; maximum time on study was 28 months.
Population: Efficacy analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 23 | 27
Months | 13.2 [4.4 to NA] — Could not be estimated due to insufficient number of events | 13.3 [4.9 to NA] — Could not be estimated due to insufficient number of events

9. Secondary Outcome: Serum Concentration of Ociperlimab
Time Frame: Predose and end of infusion (EOI) on Cycle 1 Day 1 (C1D1), Cycle 2 Day 1, Cycle 5 Day 1, Cycle 9 Day 1, and Cycle 17 Day 1
Population: Pharmacokinetic (PK) analysis set includes all participants who received any dose of study drug(s), for whom any quantifiable postdose PK concentrations were available. Results are reported for participants with available data at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 24 | 29
μg/mL
  Predose C1D1 | NA (NA) — Could not be estimated as no participants with measurable concentrations. | NA (NA) — Could not be estimated as no participants with measurable concentrations.
  EOI C1D1: number analyzed (Participants) | 24 | 27
  EOI C1D1 | 323.96 (21.810) | 296.48 (18.832)
  Predose C2D1: number analyzed (Participants) | 18 | 21
  Predose C2D1 | 61.84 (36.832) | 63.68 (38.413)
  EOI C2D1: number analyzed (Participants) | 3 | 4
  EOI C2D1 | 371.62 (24.589) | 389.27 (18.555)
  Predose C5D1: number analyzed (Participants) | 5 | 5
  Predose C5D1 | 127.20 (45.138) | 184.09 (27.675)
  EOI C5D1: number analyzed (Participants) | 5 | 6
  EOI C5D1 | 450.52 (10.707) | 507.48 (15.295)
  Predose C9D1: number analyzed (Participants) | 4 | 4
  Predose C9D1 | 181.58 (46.927) | 184.83 (23.101)
  Predose C17D1: number analyzed (Participants) | 1 | 0
  Predose C17D1 | 320.00 |

10. Secondary Outcome: Host Immunogenicity: Number of Participants With Anti-drug Antibodies (ADA) to Ociperlimab
Description: The number of participants with anti-drug antibodies to ociperlimab includes participants that were ADA-negative at Baseline and ADA-positive after drug administration during the treatment or follow-up observation period and participants who were positive at Baseline for ADA and with significant increases (4-fold or higher) in ADA titer after drug administration during the treatment or follow-up observation period.
Time Frame: From first dose of study treatment to 30 days after last dose; maximum time on treatment was 98 weeks
Population: The Immunogenicity Analysis Set is defined as all participants who received any dose of any study drug(s), for whom both Baseline ADA and ≥ 1 postbaseline ADA results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
Number analyzed (Participants) | 19 | 24
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from enrollment through the end of the study, maximum time on study was 28 months. Adverse events were assessed from first dose of study treatment to 30 days after last dose; maximum time on treatment was 98 weeks.
Groups:
- Ociperlimab + Rituximab: Participants received ociperlimab 900 mg and rituximab 375 mg/m2 Q3W by intravenous injection until confirmed progressive disease, death, withdrawal of consent, loss of follow-up, or the end of study.
Arm/Group | Ociperlimab + Tislelizumab | Ociperlimab + Rituximab
All-Cause Mortality (participants affected / at risk) | 13/24 | 14/29
Serious Adverse Events (participants affected / at risk) | 9/24 | 8/29
Other Adverse Events (participants affected / at risk) | 23/24 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ociperlimab + Tislelizumab (N=24) | Ociperlimab + Rituximab (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Death (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (3) | 0 (0)
Oral infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (3) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Shock (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ociperlimab + Tislelizumab (N=24) | Ociperlimab + Rituximab (N=29)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 8 (12)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (7)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Ocular toxicity (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 2 (3)
Fatigue (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (6) | 4 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 3 (7)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 3 (3) | 1 (1)
Apolipoprotein B increased (Investigations) | 0 (0) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 4 (5)
Bile acids increased (Investigations) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (4) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 1 (6) | 2 (3)
Blood glucose increased (Investigations) | 0 (0) | 1 (2)
Blood immunoglobulin A decreased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
Blood immunoglobulin M decreased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 5 (7) | 6 (8)
Blood pressure increased (Investigations) | 2 (4) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2)
Cystatin C increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 1 (1)
Globulins decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (10) | 5 (14)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (10) | 9 (31)
Neutrophil count increased (Investigations) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 7 (7)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 1 (1)
Serum amyloid A protein increased (Investigations) | 0 (0) | 2 (3)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 7 (11) | 7 (26)
White blood cell count increased (Investigations) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (5) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (7) | 2 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Poor quality sleep (Psychiatric disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (12)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Inadequate diet (Social circumstances) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT05267054/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT05267054/SAP_001.pdf